CLINICAL TRIAL: NCT00958373
Title: Risk Factors for Psychiatric Disorders Associated With Adolescent Idiopathic Scoliosis
Status: Withdrawn | Type: Observational
Why Stopped: Didn't have the resources necessary to carry out the study
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H08-02333
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2011-06

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; adolescent idiopathic scoliosis; spine curve; pediatric; mental health; screening
MeSH Terms: conditions — Scoliosis; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this pilot study is to determine the presence, frequency, and severity of mental health disorders amongst adolescents undergoing spinal surgery for scoliosis.

DETAILED DESCRIPTION:
This study is a cross-sectional pilot study investigating the prevalence of psychiatric illness at various time points in the course of treatment of AIS. Three independent sets of questionnaires will be administered during a single scheduled clinical visit. There will be no clinical visits for the exclusive purpose of completing questionnaires. The first questionnaire will be the SRS outcome instrument. The second questionnaire will be the Achenbach YSR, completed by the adolescents, and the parents will be asked to complete the CBCL. Finally, a generic outcome measure specific to children and adolescents, the Pediatric Outcome Data Collection Instrument, will be administered. The time requirement to complete these questionnaires is anticipated to be approximately 45 minutes. The Achenbach questionnaires will be scored promptly after each is completed using the provided scoring templates. This data will be used to identify those at risk and make appropriate resources available. This would provide appropriate care for adolescents at high risk of mental health disorder by identifying those at risk via a non-invasive screening tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AIS between the ages of eleven and sixteen, scheduled to undergo surgical intervention
* The patient and one parent will be required to complete the questionnaires in their entirety at the predetermined time points.
* There are several different methods of surgical intervention for AIS, however there will be no selection on the basis of the type of intervention.
* Curve pattern and severity will, similarly, not be used as inclusion criteria.

Exclusion Criteria:

* All types of scoliosis besides AIS will be excluded. This includes neuromuscular, congenital, infantile idiopathic, and childhood idiopathic scoliosis.
* Children younger than eleven years or older than sixteen years will be excluded.
* Those with additional chronic disease will be excluded, due to the possibility of confounding.
* Those unable to complete the entire questionnaire, for any reason, or those unable to complete the questionnaires at each time point will be excluded.
* Existence of psychiatric disorder prior to treatment will not be cause for exclusion from the study.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients between the ages of eleven and sixteen who may have a prevalence of psychiatric illness at various time points in the course of treatment of AIS.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Reilly, Dr., Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital Department of Orthopaedics, Vancouver, British Columbia, Canada